CLINICAL TRIAL: NCT01715571
Title: Clinical and Physiological Assessment of Noninvasive Penile Afferent Vibratory Stimulation of Both Surfaces of the Penis Using the Viberect® Device in Men With Mild to Moderate ED
Brief Title: Assessment of Penile Vibratory Stimulation Using the Viberect in Men With Mild-Moderate ED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain adequate recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00130002
Record Dates: First submitted 2012-10-21; First posted 2012-10-29 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Organic Erectile Dysfunction
Keywords: erectile dysfunction; vibratory stimulation; viberect
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Viberect treatment (Experimental): Participants in this arm have documented mild to moderate ED of organic etiology and will be given the Viberect device for 4 weeks of daily home use in preparation for sexual activity. Men will be asked to use the device and attempt sexual intercourse at least 3 times weekly
  Interventions: Device: Viberect

INTERVENTIONS:
Device: Viberect — Men will be asked to perform vibratory stimulation of the penis in the privacy of their home, while focused on sexual thoughts for approximately 7-10 minutes (depending on erectile response) for 3 times a week, one day apart, throughout the four week period. Men can perform the stimulation once daily, as long as each session is more than 24 hours apart.
  Men will record device use and intercourse attempts after device use in a diary.

SUMMARY:
The primary objective of this study is to assess the safety, acceptability, and satisfaction of penile vibratory stimulation in treatment of erectile dysfunction (ED). The secondary objective is to demonstrate subjective physiological response (erection, rigidity, orgasm) after four weeks of frequent device use and the satisfaction of penile erection and sexual intercourse with partner.

DETAILED DESCRIPTION:
ED is the inability to develop and maintain an erection for satisfactory sexual intercourse or activity. ED is a highly prevalent medical condition often associated with multiple causes. It is estimated that more than 50 million American men suffer from mild/moderate to severe ED. Roughly 50% of men in their 50's, 60% of men in their 60's, and 70% of men in their 70's suffer from ED. The economic impact of ED is in the billions of dollars. More than 5 billion dollars a year are spent on the pro-erectile medications currently in the market.

Penile vibratory stimulation mimics rapid and repetitive manual/hand stimulation of the penis. Vibratory stimulation of genitalia is considered safe by the medical community with important benefits including treatment of orgasmic dysfunction and stress urinary incontinence. No significant physical or emotional side-effects have been reported in the medical literature. A recent epidemiological study of the use of vibrators by American women and men has shown no complaints, and generally high satisfaction and improvement in sexual response.

Penile erection is controlled by spinal autonomic centers, the activity of which is dependent on input from supraspinal centers and the genitalia. From a neurophysiological viewpoint, scientists believe that penile erection is a culmination of multiple successful nerve reflexes that initiate a vascular event. Simultaneous vibratory stimulation of both surfaces of the penis at high frequency (70-110 Hz) for 7-10 minutes can lead to gradual filling of the penis with arterial blood within minutes by activating the pudendo-cavernosal reflex. Additional physiological effects include progressive rhythmic contraction of the perineal muscles via the bulbocavernosus reflex, which helps in strengthening rigidity of erection. This will prepare the user for successful sexual intercourse. Subsequent orgasm and ejaculation can be very strong and amplified due to stronger contraction of the bulbospongiosus muscle and activation of higher ejaculatory centers.

This study will assess daily or on-demand ease of use, safety, satisfaction, and efficacy of the home use of the Food and Drug Administration (FDA) cleared Viberect device by men with mild to moderate ED

ELIGIBILITY:
Inclusion Criteria

* mild-moderate erectile dysfunction based on International Index of Erectile Function (IIEF) erectile function score 13-25

Exclusion Criteria

* Men with neurological disease
* IIEF score less than 13
* Spinal cord injury
* History of priapism
* Pelvic neuropathy
* Post-prostatectomy
* Penile skin lesions or ulcers
* Inability to understand and demonstrate device use instructions

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Frederick Urology Specialists, Frederick, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Viberect Treatment: Single-center, non-randomized, single-arm study The Viberect device was used for 7-10 minutes at least 3 times each week, at least 24 hours apart, 4 weeks period
Period: Overall Study
Arm/Group | Viberect Treatment
Started | 11
Completed | 3
Not Completed | 8
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Groups:
- Viberect Treatment: Single-center, non-randomized, single-arm study Participants received Viberect treatment for 4 weeks of daily home use in preparation for sexual activity
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Ease/Acceptability of Use of the Viberect as Assessed by EDITS Questionnaire
Description: The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire will be administered. This is an 11 item tool addressing participant satisfaction with the Viberect. Each item is a 5-point Likert-type scale from 0 "no satisfaction or dissatisfaction" to 4 "high satisfaction." Total scoring ranges from 0-44 with higher scores indicating higher treatment satisfaction.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 21.3 (16.1)

2. Primary Outcome: Acceptability of Use of the Viberect as Assessed by TSS
Description: The Treatment Satisfaction Scale (TSS) questionnaire (patient baseline module) will be administered addressing participant satisfaction before Viberect treatment; This is an 8 item tool and each item is a 5-point Likert-type scale from 1 to 5. The score range for TSS is 8-40 with higher scores indicating greater dissatisfaction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 25 (6.1)

3. Primary Outcome: Assessment of Ease/Acceptability of Use of the Viberect as Assessed by EDITS Questionnaire
Description: as for outcome 1
Time Frame: Week 4
Population: Patient 1 data is missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 2
score on a scale | 15 (12.7)

4. Primary Outcome: Acceptability of Use of the Viberect as Assessed by TSS
Description: The Treatment Satisfaction Scale (TSS) questionnaire (patient active treatment module) will be administered addressing participant satisfaction following Viberect treatment; This is a 13 item tool and each item is a 5-point Likert-type scale from 1 to 5. The score range for TSS is 13-65 with higher scores indicating greater dissatisfaction.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 38.3 (16.1)

5. Secondary Outcome: Erectile Function (EF) as Assessed by the International Index for Erectile Function (IIEF)-5 Questionnaire
Description: The International Index for Erectile Function (IIEF)-5 questionnaire will be administered. This is a 5 item tool; addressing Erectile function over the previous 4 weeks. Scores from 1-25 can be obtained in this domain. Scores are interpreted as follows: 1-7 = Severe Erectile dysfunction (ED), 8-11 = Moderate ED, 12-16 = mild-moderate ED, 17-21 = mild ED, 22-25 = No ED
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 14.6 (1.15)

6. Secondary Outcome: EF as Assessed by the Erectile Hardness Score (EHS)
Description: The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single-item tool. It is scored from 1 to 4. Higher scores indicate better erection rigidity.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 2.33 (0.5)

7. Secondary Outcome: EF as Assessed by the International Index for Erectile Function (IIEF)-5 Questionnaire
Description: as for outcome 5
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 16.3 (1.52)

8. Secondary Outcome: EF as Assessed by the Erectile Hardness Score (EHS)
Description: as for outcome 6
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Viberect Treatment
Number analyzed (Participants) | 3
score on a scale | 2.66 (0.5)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Viberect Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Among the limitations of this study are the small number of subjects, short duration of therapy, and a single-arm design with no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT01715571/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT01715571/SAP_001.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT01715571/ICF_002.pdf